CLINICAL TRIAL: NCT01065974
Title: A Test of Nutritional Interventions to Enhance Weight Loss Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Michael Lowe, Professor, Drexel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01DK80909-2; 5R01DK080909 (NIH)
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Overweight; Obesity; Weight Loss Maintenance
Keywords: Nutritional Intake; Psychosocial Outcome
MeSH Terms: conditions — Overweight; Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Behavior Therapy (Active Comparator): Behavioral treatment strategies will be utilized to facilitate adherence to the treatment goals in all three treatments. Participants in the BT condition will receive only the BT intervention. Strategies that will be emphasized are listed below:
  * Self monitoring
  * Stimulus control
  * Changing eating behaviors
  * Goal setting
  * Problem solving
  * Social support
  * Cognitive restructuring
  * Relapse prevention
  Interventions: Behavioral: Behavior Therapy
- Behavior Therapy + Meal Replacements (Experimental): The BT +MR condition will implement behavioral treatment strategies in a way that is nearly identical to that of the BT condition. However, participants in this condition also will use MRs during weight loss and weight loss maintenance.
  Interventions: Dietary Supplement: Meal Replacements
- Nutritrol (Experimental): Participants in this condition will be informed about the evidence indicating that the availability, structure and composition of foods they encounter or seek out in their daily lives will play a major role in determining their ability to maintain the weight they lose. We will present the treatment as an opportunity to make numerous changes to their "personal food environment" involving the variety, energy density, nutritional composition, and portion size of the foods they encounter in every day life.
  The Nutritrol condition is comprised of several components:
  * Food structure
  * Energy density
  * Reduce variety of foods high in energy density and increase variety of foods low in energy density
  * Protein intake
  * Controlling the personal food environment
  * Individualized weight loss maintenance prescriptions
  Interventions: Behavioral: Nutritrol

INTERVENTIONS:
Behavioral: Behavior Therapy — Weight loss using CBT and continued CBT during weight loss maintenance.
  Arms: Behavior Therapy
Dietary Supplement: Meal Replacements — Weight loss using CBT and meal replacements.
  Arms: Behavior Therapy + Meal Replacements
Behavioral: Nutritrol — To make widespread nutritional changes to participants personal food environments.
  Arms: Nutritrol

SUMMARY:
The purpose of this study is to compare standard Behavior Therapy (BT), BT plus Meal Replacements (MR) and a condition focusing on the nutritional changes to the home food environment (HFE) on weight loss, weight loss maintenance, nutritional composition of the diet and psychosocial outcomes. A second aim is to determine the degree to which the specific targets of the experimental interventions do in fact change in the anticipated direction during the intervention and to evaluate whether such changes might account for improvements in weight loss maintenance. This study is important because it could provide the first evidence that the current standard of care for obesity lifestyle treatment could be improved by the addition of MRs or a program of comprehensive nutritional change.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the ages of 18 and 65
* body mass index (BMI; kg/m2) between 27-45
* able to travel regularly to the study location
* interested in participating in a weight loss program.

Exclusion Criteria:

* currently enrolled in another organized weight loss program
* lactose intolerance
* taking medications that affect appetite (unless dosage had been stable for at least the previous six months)
* history of gastric bypass or other surgical weight loss procedures
* medical conditions (e.g., cancer, substance abuse, psychotic disorders) that could limit their ability to comply with the behavioral recommendations or pose a risk to the participant during weight loss
* pregnancy or planning to become pregnant during the next two years -
* breastfeeding
* consuming an amount of alcohol that could interfere with study completion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2009-10; Primary Completion 2016-04-30 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Body weight over time. | Baseline, 6 months, 12 months, 18 months, 24 months, 36 months
  Change in body weight measured on electronic scale.

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Lowe, Ph.D., Principal Investigator — Drexel University
Locations (2):
- United States (2):
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Lowe MR, Butryn ML, Zhang F. Evaluation of meal replacements and a home food environment intervention for long-term weight loss: a randomized controlled trial. Am J Clin Nutr. 2018 Jan 1;107(1):12-19. doi: 10.1093/ajcn/nqx005. PMID 29381791
- [Derived] Feig EH, Lowe MR. Variability in Weight Change Early in Behavioral Weight Loss Treatment: Theoretical and Clinical Implications. Obesity (Silver Spring). 2017 Sep;25(9):1509-1515. doi: 10.1002/oby.21925. PMID 28845608